CLINICAL TRIAL: NCT00874484
Title: Enoxaparin as Treatment for Vulvar Vestibulitis Syndrome - Vulvodynia
Brief Title: Enoxaparin as Treatment for Vulvodynia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Prof. Jacob Bornstein, Chair, Dpt Obstetrics & Gynecology, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JB 2409
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Clexane (enoxaparin)
- 2 (Placebo Comparator)
  Interventions: Drug: Clexane (enoxaparin)

INTERVENTIONS:
Drug: Clexane (enoxaparin) — One arm receives enoxoparin, second arm receives saline

SUMMARY:
The investigators hypothesize that injections of Low molecular weight heparin (LMWH) [enoxaparin] will reduce pain in women with vulvodynia.

ELIGIBILITY:
Inclusion Criteria:

* women with vulvodynia

Exclusion Criteria:

* women without vulvodynia

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
vestibular pain | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital- Nahariya, Nahariya, Israel

REFERENCES:
- [Derived] Farajun Y, Zarfati D, Abramov L, Livoff A, Bornstein J. Enoxaparin treatment for vulvodynia: a randomized controlled trial. Obstet Gynecol. 2012 Sep;120(3):565-72. doi: 10.1097/AOG.0b013e3182657de6. PMID 22914465